CLINICAL TRIAL: NCT02818101
Title: Hypnosis Efficacy for the Prevention of Anxiety During a Coronary Angiography
Acronym: HypCor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-02-CHRMT
Record Dates: First submitted 2016-03-30; First posted 2016-06-29 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2016-03

CONDITIONS: Coronary Angiography

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No hypnosis session before the coronary angiography
- Hypnotised group (Experimental): Hypnosis session before the coronary angiography
  Interventions: Behavioral: Hypnosis session

INTERVENTIONS:
Behavioral: Hypnosis session
  Arms: Hypnotised group

SUMMARY:
The purpose of this study is to confirm the utility for hypnosis in the coronary angiographic examination. The technique would be an alternative to prevent the consumption of anesthesic drugs.

DETAILED DESCRIPTION:
The coronary angiography is a medical imaging acquisition used in cardiology to highlight the coronary arteries after a coronary disease suspicion. According to an expert consensus it is performed under local anesthesia. Indeed the examination is quite painless, apart from the initial arterial puncture. Moreover, any patient chest pain must be detected during the examination to locate the guilty coronary injury. This is not possible with a patient under general anesthesia.

But, no general anesthesia may be a source of anxiety for patients, and the technique can be painful at several times: during the puncture, the exploration of probe into the winding, spastic or over-calcified arteries, or even during the dilation by the balloon swelling which obstructs downstream the artery.

The efficiency evaluation of the hypnosis made by INSERM in 2015 concludes that "the use of hypnosis during a surgical practice or during a medical or a interventional radiological act allows to reduce the consumption of sedative drugs and/or pain medication preoperatively".

The study hypothesis, is that hypnosis can contribute to a decreasing of anxiety and the pain for patients undergoing coronary angiography, and even a decreasing of complications due to a better control of hemodynamic (heart rate and blood pressure).

It could entail a better comfort for operator during the coronary angiography.

Primary objective :

To compare the initial anxiety state before the coronary angiographic performing scheduled for adults with no earlier coronary angiography, according to they will undergo a hypnotic session or not before the examination, with posthypnotic suggestions of self-hypnosis to make during the coronary angiography.

Secondary objective :

To compare between the two groups of patients:

* pain during and after the coronary angiography
* hemodynamic factors heart rate, blood pressure before and after the examination
* operator comfort
* use of sedative drugs, pain medication and local anesthesia
* outbreak of major and minor complications

Primary endpoint :

Anxiety measured using self-report questionnaire (STAI-Y-A ), before coronary angiography

Secondary endpoints :

Trait anxiety (STAI-Y-B questionnaire) State anxiety the eve of coronary angiography Pain before and during the coronary angiography : Visual Analog Scale (VAS) Heart rate and blood pressure before and after the coronary angiography Comfort for the operator of the angiography : Likert scale into 5 points (1 : the worst comfort, 5 : the best possible comfort) Dose of sedative drugs, pain medication and local anesthesia injected during the coronary angiography Outbreak of major complications during the coronary angiography (death, stroke, tamponade, hemorrhagic shock, anaphylactic shock against the imaging tracer, ventricular tachycardia or ventricular fibrillation, severe bradycardia) or minor complications (vagal reaction, hematoma at the puncture point, skin allergy)

Methodology :

Efficiency comparative study, randomized, simple-blind (angiography operator in blind), single center, routine clinical care Only one medical check per patient

Procedures :

When a patient is taken over in cardiology department the eve of a scheduled coronary angiography, the cardiologist purposes them to take part in this study.

If they accept, a first evaluation of anxiety (trait and state) is performed. The following day, before going to the coronary angiography room, the patients are splitted randomly into two groups :

* A group of patients which undergo a hypnotic session before examination with posthypnotic suggestions of self-hypnosis to be performed during the angiography. A medical prescription for anxiolytics can be made according to the patient clinical signs of anxiety
* Another group becomes only a prescription of anxiolytics according to the patient clinical signs of anxiety.

The State Anxiety is measured after the setting of the patient in the coronary angiography room, before performing the examination. The pain and the hemodynamic factors are measured during and after the coronary angiography. The comfort of operator is evaluated too.

The patients will be contacted by phone one month after the coronary angiography to evaluate their satisfaction with their medical care.

Patients number :

Assuming that the control group has a mean score of 50 (standard deviation 10) with STAI-Y A, and a clinically significant difference (from 5 points), 85 patients must be included in each group, so totally 170 patients.

Trial Duration :

Expected study start: first semester of 2016 Inclusion duration: 12 months Duration per patient: 1 mois Total study duration: 18 months (including the data analysis et the report of results)

Statistical Analysis:

* Primary objective: comparison of the mean scores STAI-Y A between the two groups (T test of Student), with adjustment on the potential factors of confusion (multiple linear regression)
* Secondary objective: comparison of the quantitative criteria (T tests of Student) and qualitative criteria (Fischer's exact test) between the two groups.

Expected Benefits :

Since coronary angiography is an invasive procedure without general anesthesia affecting a noble organ, this procedure could be anxiogenic and even psychologically traumatic emergency. Not practice under general anesthesia prevents potential risks for the patient, but anxiety, non-comfort and pain are existing. We think that hypnosis could improve the patient care psychologically and physically and for any invasive procedure.

In this case, fewer or no sedative drugs and pain medication will be necessary, and it would decrease their potential iatrogenesis, the patient care will be improved. It will be an alternative for patient to decrease their drugs consumption.

Quality Assurance Plan :

Data will be recorded in a Paper Case Report from medical records. The patients will undergo only one medical examination for the study. No follow-up is expected.

ELIGIBILITY:
Inclusion Criteria:

* adult
* coronary angiography scheduled with or without stenting
* registered with a social security scheme
* people informed clearly by the investigator

Exclusion Criteria:

* coronary angiography already performed
* not well french speaking and understanding
* with functional disabilities (mental disorder, ...)
* known background of schizophrenia
* deaf or hard of hearing
* patient under legally protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
State Anxiety | 1 day
  Spielberger State-Trait Anxiety Inventory (STAI):

SECONDARY OUTCOMES:
Comfort for the operator of the angiography | 1 day
  Likert scale into 5 points
Pain | 1 day
  visual analogue pain scale
Heart rate | 1 day
  beats per minute (bpm)
Blood pressure | 1 day
  mmHg
Major complications | 1 day
  beats per minutes
dose of sedative drugs | 1 day
  mg

CONTACTS AND LOCATIONS:
Locations (1):
- Chr Metz Thionville, Metz, France

REFERENCES:
- [Derived] Abensur Vuillaume L, Gentilhomme C, Weber S, Ouamara N, Bayard J, Valla M, Khalife K, Goetz C, Guler N. Effectiveness of Hypnosis for the Prevention of Anxiety During Coronary Angiography (HYPCOR study): a prospective randomized study. BMC Complement Med Ther. 2022 Nov 29;22(1):315. doi: 10.1186/s12906-022-03792-x. PMID 36447198